CLINICAL TRIAL: NCT05992961
Title: The Effects of Troponin I Surveillance Among Patients Undergoing Acute High-risk Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P-2020-507-2
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Abdomen, Acute; Myocardial Injury After Non-cardiac Surgery; Troponin I; Myocardial Injury; Emergency Surgery
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients not undergoing troponin I surveillance: Patients undergoing acute high-risk abdominal surgery during the period February 1, 2018, to February 28, 2019. No troponin I measurements were made.
- Patients undergoing troponin I surveillance: Patients undergoing acute high-risk abdominal surgery during the period March 1, 2019, to February 28, 2021 as well as postoperative troponin I surveillance .
  Interventions: Diagnostic Test: Troponin I

INTERVENTIONS:
Diagnostic Test: Troponin I — Troponin I were measured 6-12 hours postoperatively and on each of the succeeding four postoperative days for patients operated March 1, 2019, to February 28, 2021.
  Patients with increased troponin I levels were assessed regarding symptoms of myocardial ischaemia including electrocardiography. Each patient was individually assessed, and relevant treatment and follow-up were planned in collaboration between surgeons, cardiologists, and anaesthesiologists.
  Groups: Patients undergoing troponin I surveillance

SUMMARY:
Treatment of disorders such as gastrointestinal tract (GI) perforation, ischemia and obstruction often require acute high-risk abdominal surgery, which is associated with a high risk of complications such as myocardial injury after non-cardiac surgery (MINS) and mortality. The majority of patients with MINS will not experience any symptoms, and thus MINS remains undetected without routine troponin measurements.

The investigators hypothesized that implementing surveillance with troponin I as a standard care might be useful as risk stratification, and that increased surveillance, examinations, and subsequent individually based medical interventions, might improve the outcomes for patients with MINS.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were 18 years or older
* Undergoing surgery for gastrointestinal perforation, obstruction, mesenterial ischemia or necrosis, or anastomotic leakage.

Exclusion Criteria:

* Not undergoing surgery for one of the conditions above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing acute high-risk abdominal surgery at Copenhagen University Hospital - North Zealand, Denmark during the period February 1, 2018, to February 28, 2021.
  For patients undergoing acute high-risk abdominal surgery on more than occasion during the period of observation, only the first case of surgery was included.
Sampling Method: Probability Sample
Enrollment: 558 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
compare the mortality rate before and after implementing troponin I surveillance | 30-, 90-, and 365-day
  compare the 30-, 90-, and 365-day mortality rate after acute hugh-risk abdominal surgery in patients undergoing postoperative troponin I surveillance and subsequent intervention with a historical group of patients not undergoing troponin I surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Anders TB Bertelsen, PhD, MD, Principal Investigator — Copenhagen University Hospital - North Zealand
Locations (1):
- Copenhagen University Hospital - North Zealand, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD can be shared at request.